CLINICAL TRIAL: NCT06306079
Title: The Possibilities and Acceptability of Applying Gait Modification to the Treatment of Knee Osteoarthritis in Saudi Arabia Based on the Perceptions of Patients and Physiotherapists. A Mixed-methods Feasibility Study.
Brief Title: Using Gait Modification to Treat Knee Osteoarthritis in Saudi Arabia: Possibilities and Acceptability.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Khalid University (Other)
Collaborators: University of Nottingham (Other)
Responsible Party: Principal Investigator, Abdullah Al Assiri, Principal Investigator, King Khalid University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KKUMC; Abdullah Al Assiri (Other: King Khalid University Medical City); Prof Pip Logan (Other: Professor of Rehabilitation Research, University of Nottingham, UK.); Professor Ana Valdes (Other: Professor of Molecular & Genetic Epidemiology, University of Nottingham, UK.); Dr. Benjamin Smith (Other: Doctor of Physiotherapy, Division of Rehabilitation and Ageing, University of Nottingham. UK.)
Record Dates: First submitted 2022-12-31; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Osteoarthritis, Knee; Pain; Biomechanical Lesion
Keywords: Knee osteoarthritis; Insole; Biomechanical; Saudi Arabia
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Intervention Model Description: A gait modification (Lateral wedge insole) program will be conducted over 4 to 6 weeks in the physiotherapy gym or adjusted treadmill and outside the clinic during the day (at least 8 hours per day).
  * During the session, the researcher will observe participants inside the clinic and ensure that the modified gait application is applied, and outside the clinic will be followed by telephone.
  * Participants will walk on the gym floor or an adjusted treadmill for at least 15 to 20 minutes during each session. Participants will be instructed to use the mirror for feedback and achieve the target modified gait procedure. However, it will be emphasised gait modification procedures exhibited at baseline pain and function, and then at the end of the trial, it will focus on subjects' acceptability.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility intervention (Experimental): The intervention will be foot insole (lateral wedge) insole, which has already been delivered in routine UK NHS and SA environments by at least one physiotherapist. Clinical testing will be done with 15-25 knee osteoarthritis subjects. These individuals will be assigned to a single intervention group for 4-6 weeks of re-gait training intervention. It involves a personalised gait retraining programme (sizable insole) for the KOA subjects to evaluate the impact on knee pain and improve function. It is set within 4-6 weeks of VAS and the WOMAC tools for knee pain & function outcome.
  Interventions: Device: Lateral Wedge insole

INTERVENTIONS:
Device: Lateral Wedge insole — Insoles with lateral wedges are placed in patients' shoes to control biomechanical knee loading on the medial side of the knee. Insoles with lateral wedges are designed to be thinner on the inside (medially of the foot) and thicker on the outside (laterally of the foot) to relieve knee biomechanical loading parameters.
  Other Names: Footwear insole; Ankle foot orthoses

SUMMARY:
A variety of biomechanical gait modification interventions can elevate knee loading and improve knee symptoms in knee osteoarthritis patients. However, there was a lack of acceptability and adherence regarding modification interventions without any explanation.

Thus, this study investigates the feasibility and acceptability of foot insoles as a gait modification tool among Saudi Arabian knee osteoarthritis patients and physiotherapists.

This study aims to answer the following:

* Which gait modification intervention is most likely to be implemented in Saudi Arabia (SA) clinical practice, taking context, patients' clinical and research evidence into consideration?
* In Saudi Arabia, can this proposed foot-insole intervention be implemented? Is there sufficient experience among physiotherapists regarding gait modification to deliver it, and will patients engage with it? How can KOA rehabilitation outcomes be evaluated in the future?

The participants will be conducted over three phases:

1. The patients' interview and therapists' focus group discussion will be used to examine KOA patients' and clinicians' perspectives on enabling and accepting gait modifications in phase 1.
2. The feasibility study will explore how a small number of KOA patients tolerate gait modifications and consider the most relevant outcome measures, such as pain and function, in phase (2).
3. A small group of knee osteoarthritis patients and their physiotherapists who participated in phase (2) will be asked to participate in a descriptive survey in phase (3). To examine the acceptability and feasibility of the study intervention in phase (2).

DETAILED DESCRIPTION:
Since several different types of gait modifications have been studied, it has been challenging to determine which are most likely to be used by patients and healthcare professionals.

A notable number of Saudi Arabians suffer from knee osteoarthritis (KOA), which reported a 29.5% prevalence of KOA; another recent study reported a 24.5% prevalence of KOA among the elderly. A 2002 study found that 30.8% of those aged 46-55 and 60.6% aged 66-75 were affected. Thus, KOA is roughly equally distributed between genders and is more prevalent among elderly and overweight individuals, so policymakers should focus on raising awareness to prevent and treat affected individuals. The healthcare system in SA is publicly funded and accessible; 79% of patients use the public system, and the rest obtain private care. In most cases, private patients have insurance coverage. The public healthcare system has three primary, secondary, and tertiary care levels. Rehabilitation and gait modification investigations are not available at the primary level.

This snapshot of the literary review raises questions about the viability of the long-term use of learned/assistive gait modifications. The studies reported dissatisfaction with the gait modification approach but gave no reasons. Since most studies focus on results in a short time or a specific area, pre-training courses measuring acceptability and commitment can fill the gaps in previous studies. After determining the importance of gait modification, the question becomes, should it be integrated into the therapy strategy or other rehabilitative methods to increase the treatment's clinical efficacy? It is essential to understand the practices, views and expectations of KOA patients and health professionals concerning gait modifications.

ELIGIBILITY:
Inclusion Criteria:

KOA Patient participants:

* Adults aged above 45 years old.
* Both Male & Female.
* Radiographically or KOA participants meet any diagnostic classification guidelines/criteria (American College of Rheumatology classification criteria) or any eligible diagnostic guidelines.
* Typical knee pain while walking > 3 on an 11-point scale (0-10) in at least one knee pain or tenderness, primarily in the medial knee.

Exclusion Criteria:

* Severe KOA subjects (on the waiting list for knee arthroplasty).
* Knee post-operation or corticosteroid intra-articular injection last 6 months.
* Inability to walk for longer than 20 minutes without experiencing severe pain.
* Painful treadmill walking or unable to walk without heavy assistance, such as a lifting belt or walker frame.
* Significant knee effusion, musculoskeletal or neurological diseases that influence gait parameters.
* It is presently undergoing physiotherapy treatment.
* Rheumatoid Arthritis (RA), gout, one or both knees replaced, low back pain, hip OA, any serious knee or lower limb injuries in the past 24 months.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Pain level | 6 weeks post-intervention.
  The change from baseline pain intensity level at 6-weeks, based on the nine points of a visual analogue scale, where 0 represents (no pain) and 9 represents (worst pain).
Western Ontario and McMaster Universities Arthritis Index-total | 6 weeks post-intervention.
  The change from baseline pain, stiffness and physical activity levels at 6-weeks.
  Each question is scored from 0 to 4, which are: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4).
  Scores are summed for each subscale, ranging from 0-20 for pain, 0-8 for stiffness, and 0-68 for Physical Function.
  A higher WOMAC score indicates worse pain, stiffness, and functional limitations.
Likert scale | 6 weeks post-intervention.
  Measuring knee osteoarthritic subjects' satisfaction based on the 5 point Likert scale survey.
Likert scale | 6 weeks post-intervention supervision.
  Measuring therapists' agreement based on the 5-point Likert scale survey.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Al Assiri, PhD student, Principal Investigator — University of Nottingham
Locations (1):
- King Faisal Specialist Hospital & Research Centre, Jeddah, Western, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Al-Arfaj A, Al-Boukai AA. Prevalence of radiographic knee osteoarthritis in Saudi Arabia. Clin Rheumatol. 2002 May;21(2):142-5. doi: 10.1007/s10067-002-8273-8. PMID 12086165
- [Result] Al-Modeer MA, Hassanien NS, Jabloun CM. Profile of morbidity among elderly at home health care service in Southern Saudi Arabia. J Family Community Med. 2013 Jan;20(1):53-7. doi: 10.4103/2230-8229.108187. PMID 23723732
- [Result] Khalid W. AlKuwaity, Tasneem N. Mohammad, Malik A. Hussain, Annas Alkhanani, A. M. . A. (2018) 'Prevalence and Determinant Factors of Osteoarthritis of the Knee Joint among Elderly in Arar, KSA', The Egyptian Journal of Hospital Medicine, 72(9).
- [Result] Almalki M, Fitzgerald G, Clark M. Health care system in Saudi Arabia: an overview. East Mediterr Health J. 2011 Oct;17(10):784-93. doi: 10.26719/2011.17.10.784. PMID 22256414
- [Result] Pollo FE, Otis JC, Backus SI, Warren RF, Wickiewicz TL. Reduction of medial compartment loads with valgus bracing of the osteoarthritic knee. Am J Sports Med. 2002 May-Jun;30(3):414-21. doi: 10.1177/03635465020300031801. PMID 12016084
- [Result] Butler RJ, Marchesi S, Royer T, Davis IS. The effect of a subject-specific amount of lateral wedge on knee mechanics in patients with medial knee osteoarthritis. J Orthop Res. 2007 Sep;25(9):1121-7. doi: 10.1002/jor.20423. PMID 17469197
- [Result] Kutzner I, Damm P, Heinlein B, Dymke J, Graichen F, Bergmann G. The effect of laterally wedged shoes on the loading of the medial knee compartment-in vivo measurements with instrumented knee implants. J Orthop Res. 2011 Dec;29(12):1910-5. doi: 10.1002/jor.21477. Epub 2011 Jun 8. PMID 21656850
- [Result] Fantini Pagani CH, Hinrichs M, Bruggemann GP. Kinetic and kinematic changes with the use of valgus knee brace and lateral wedge insoles in patients with medial knee osteoarthritis. J Orthop Res. 2012 Jul;30(7):1125-32. doi: 10.1002/jor.22032. Epub 2011 Dec 12. PMID 22161816
- [Result] Jones RK, Zhang M, Laxton P, Findlow AH, Liu A. The biomechanical effects of a new design of lateral wedge insole on the knee and ankle during walking. Hum Mov Sci. 2013 Aug;32(4):596-604. doi: 10.1016/j.humov.2012.12.012. Epub 2013 Jul 17. PMID 24054897
- [Result] Moyer RF, Birmingham TB, Dombroski CE, Walsh RF, Leitch KM, Jenkyn TR, Giffin JR. Combined effects of a valgus knee brace and lateral wedge foot orthotic on the external knee adduction moment in patients with varus gonarthrosis. Arch Phys Med Rehabil. 2013 Jan;94(1):103-12. doi: 10.1016/j.apmr.2012.09.004. Epub 2012 Sep 17. PMID 22995151

DOCUMENTS (1):
  • Study Protocol (2023-01-04): https://cdn.clinicaltrials.gov/large-docs/79/NCT06306079/Prot_000.pdf